CLINICAL TRIAL: NCT03193385
Title: Evaluation of Closed Reduction for Treatment of Developmental Dysplasia of the Hip in Children
Brief Title: Treatment of Developmental Dysplasia of the HIp
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Emad Abdelmaged Abdelqawi, Principal investigator, Assiut University
Other Study IDs: DDH
Record Dates: First submitted 2017-06-16; First posted 2017-06-20 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Hip Dysplasia
MeSH Terms: conditions — Hip Dislocation | interventions — Closed Fracture Reduction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Closed reduction
  Interventions: Procedure: closed reduction

INTERVENTIONS:
Procedure: closed reduction — Closed reduction is where the thigh bone is placed into the socket without any surgical incision being made. This is more likely to be performed in a child under the age of four year. The femoral head is gently manipulated into the socket, whilst the child is under anaesthetic. Once the femoral head is in place, a hip Spica is applied and can remain in place for up to three months to maintain the hip in the correct position. This allows time for healing and for the socket and the thigh bone to mould together as a joint.

SUMMARY:
Closed reduction is where the thigh bone is placed into the socket without any surgical incision being made. This is more likely to be performed in a child under the age of four year. The femoral head is gently manipulated into the socket, whilst the child is under anaesthetic. Once the femoral head is in place, a hip Spica is applied and can remain in place for up to three months to maintain the hip in the correct position. This allows time for healing and for the socket and the thigh bone to mould together as a joint.

The purpose of this study was to identify and evaluate risk factors of avascular necrosis (AVN) after closed treatment for developmental dysplasia of the hip (DDH).

assessed according to Salter's classification system.

DETAILED DESCRIPTION:
Technique of closed reduction Preoperative Patients were admitted one day before operation in the pediatric ward and when possible skin traction was applied for the affected side. Blood sample was extracted for basic lab work investigations Blood bank was contacted to prepare cross matching for blood in case of shifting the procedure to open reduction. The side of DDH was marked and patient kept fasting starting from midnight before operation.The consent was signed by the legal guardian and we included the possibility of turning closed to open reduction in case of failure to obtain concentric reduction intraoperatively Operative technique After induction of general anesthesia with proper muscle relaxant,the patient was examined gently for hip mobility and possibility of closed reduction.Vigorous maneuvers were avoided.The hip was reduced by placing it in flexion beyond 90 degrees and gradually abducting it while gently lifting the greater trochanter, as is done during the Ortolani maneuver. The minimum possible force was applied and after a palpable reduction was felt, the hip was moved to determine the range of motion in which it remained reduce as described by Ramsey and associates. The hip was adducted to the point of redislocation, and that position was noted. The hip was again reduced and then extended until it dislocates, and the point of dislocation was noted. If the hip required internal rotation to maintain reduction, this was also noted

Tenotomy

At times, an adductor tenotomy was used to increase the safe zone by allowing for a wider range of abduction. However,wide abduction should never be used because It is known that this can predispose to AVN.Excessive internal rotation is also a known cause of AVN and thus must be avoided.A percutaneous adductor tenotomy under sterile conditions was performed for mild adduction contractures. For more severe adduction contracture or one of long duration,an open adductor tenotomy through a small transverse incision was done

Technique of cast application Closed reduction of the hip should be performed under general anesthesia in the operating room to provide adequate muscle paralysis. The reduction maneuver involves longitudinal traction, flexion, and abduction of the hip, all while applying posterior pressure on the greater trochanter [12]. Frequently an adductor tenotomy is necessary via an open or percutaneous technique, which relieves one of the opposing forces and widens the "safe zone." After reduction of the hip, intraoperative arthrography will confirm a concentric reduction of the femoral head by demonstrating a collection of dye in the space between the femoral head and medial border of the acetabulum of less than 5-7 mm [13]. The previously described collection of dye is often referred to as the "medial dye pool." If the medial dye pool measures greater than 7 mm, it is an indication to proceed with an open reduction [13]. Once reduction of the hip has been documented, the stable zones of the hip in all planes of direction (abduction/adduction, flexion/extension, internal/ external rotation) should be identified to ensure stability of the hip in the "human position" prior to applying the spica cast. The purpose of the spica cast is to maintain the hip in 100 of flexion and 40-50 of abduction, which is commonly referred to as the "human position" of the hip . The spica cast is technically demanding, but close attention to detail can ensure hip positioning and maintenance of the reduction. Because the padding over the anterior aspect of the hip has a tendency to extend the hip, it is prudent to maintain necessary flexion until the casting material has hardened. The femoral head will often migrate posteriorly leading to a loss in the reduction, but the use of a greater trochanter mold can help prevent the migration .

Confirming of closed reduction by arthrography inter operative and C T /MRI post-operative

ELIGIBILITY:
Inclusion Criteria:

* Children that missed the initial diagnosis after birth and presented around six months up to four years which included in this study. All patients did not receive prior treatment such as Pavlik harness or splints.

Exclusion Criteria:

* Patients with neurological, septic, traumatic or syndromatic dislocation is not included in our study.

Ages: 6 Months to 4 Years | Sex: All
Age Groups: Child
Study Population: closed reduction of the neglected hip dyplasia The purpose of this study to identify predictive factors that would best indicate the satisfactory function and radiological outcome after close redaction of developmentlal dysplasia of the hip in children
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2017-07 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Harris Hip score | 6 month
  harris hip score for function of the hip

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anuar R, Mohd-Hisyamudin HP, Ahmad MH, Zulkiflee O. The Economic Impact of Managing Late Presentation of Developmental Dysplasia of Hip (DDH). Malays Orthop J. 2015 Nov;9(3):40-43. doi: 10.5704/MOJ.1511.006. PMID 28611908
- [Background] de Hundt M, Vlemmix F, Bais JM, Hutton EK, de Groot CJ, Mol BW, Kok M. Risk factors for developmental dysplasia of the hip: a meta-analysis. Eur J Obstet Gynecol Reprod Biol. 2012 Nov;165(1):8-17. doi: 10.1016/j.ejogrb.2012.06.030. Epub 2012 Jul 21. PMID 22824571
- [Background] Brady RJ, Dean JB, Skinner TM, Gross MT. Limb length inequality: clinical implications for assessment and intervention. J Orthop Sports Phys Ther. 2003 May;33(5):221-34. doi: 10.2519/jospt.2003.33.5.221. PMID 12774997
- [Background] Sarkissian EJ, Sankar WN, Baldwin K, Flynn JM. Is there a predilection for breech infants to demonstrate spontaneous stabilization of DDH instability? J Pediatr Orthop. 2014 Jul-Aug;34(5):509-13. doi: 10.1097/BPO.0000000000000134. PMID 24590335
- [Background] Race C, Herring JA. Congenital dislocation of the hip: an evaluation of closed reduction. J Pediatr Orthop. 1983 May;3(2):166-72. doi: 10.1097/01241398-198305000-00004. PMID 6863522